CLINICAL TRIAL: NCT06266026
Title: ThermoBreast - Non-contact Breast Cancer Imaging Using AI-enhanced Thermography. An International, Multicenter, Prospective Development and Validation Trial.
Brief Title: ThermoBreast - Non-contact Breast Cancer Imaging Using AI-enhanced Thermography.
Acronym: ThermoBreast
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ThermoMind Ltd. (Industry)
Collaborators: Assuta Medical Centers Ltd. (Unknown); Hospital of Lithuanian University of Health Sciences Kaunas Clinics (Unknown); Institut Gustav Roussy (Unknown); M.D. Anderson Cancer Center (Other); Sheba Medical Center (Other Government); Holy Family Hospital, Nazareth, Israel (Other); University College Cork (Other); Univerzitetni klinicni center Maribor (Unknown); Academisch Ziekenhuis Groningen (Other); Technical University of Munich (Other); Technion, Israel Institute of Technology (Other); Vrije Universiteit Brussel (Other); Cancer Patients Europe (Unknown); University Hospital Heidelberg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: ThermoBreast
Record Dates: First submitted 2023-11-18; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
Keywords: Artificial Intelligence; Thermography; breast imaging; breast diagnosis
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ThermoBreast - AI-based evaluation of dynamic breast thermography imaging — Index test: AI-based evaluation of dynamic breast thermography imaging (ThermoBreast). The ThermoBreast evaluation will be performed independently of the routine breast cancer diagnostic evaluation. Some baseline risk variables (e.g. patient age, hormonal status) may be included in the ThermoBreast evaluation.
  Reference test: Routine breast diagnostics will serve as a reference test against which the ThermoBreast outcome will be compared. Depending on national guidelines and clinical scenarios, routine breast cancer diagnostics can consist of several routine procedures, including clinical examination, ultrasound, mammography, tomosynthesis, MRI, follow-up imaging, biopsy, surgical excision, and histopathologic evaluation. All procedures will be performed as indicated and specified by the respective, current national guidelines.
  Other Names: ThermoMind Vision One Device

SUMMARY:
Breast cancer is one of the most worrisome health concerns facing women. Early detection and active patient monitoring are crucial to survival. The chances of a cure are high when detected and treated in the early stages. Standard breast cancer diagnostic methods such as mammography, ultrasound, and MRI have limitations such as ionizing radiation, high false-positive rates, and/or high expenses.

Medical Thermography might overcome these limitations: It is a non-invasive , adjunctive physiologic imaging technology that uses a high-resolution infrared camera and computer processing to produce an image (thermogram) of a patient's skin surface temperatures. It is a non-contact screening method, which does not involve radiation exposure or invasive procedures, and is safe for both the patient and the trained personnel performing the screening. While mammography and ultrasound depend primarily on structural and anatomical variation of the tumor from the surrounding breast tissue, thermography detects pathophysiological changes within the breast such as metabolic and vascular changes caused by cancer. The heat transfer in the body is conducted by the circulatory system; hence, pathologies identified by thermography are generally associated with changes in blood perfusion.

To date, there has been no completed or ongoing large-scale, prospective, multicenter, international study that evaluates the diagnostic performance of thermal video streams coupled with advanced Artificial Intelligence algorithms for early-stage breast cancer screening and diagnosis. The proposed study will be crucial for the development of a new imaging modality that aims to be both cost-effective and to carry a minimal level of risk, facilitating screening of women of all age groups and breast densities, enabling early detection of abnormalities caused by malignant processes and improving patient monitoring.

DETAILED DESCRIPTION:
This study is designed as a multicenter, prospective, blinded, three cohorts, diagnostic trial. Patients will be recruited at 11 centers in France, Germany, Ireland, Israel, Slovenia, Lithuania, and the US.

The primary objective is to compare the diagnostic performance of advanced image processing AI models to automatically predict breast malignancy based on thermograms and individual patient data collected during breast examination (ThermoBreast) with routine breast cancer screening and imaging.

The study population consists of women undergoing routine screening for breast cancer or diagnostic evaluation of suspicious breast masses. The study will recruit women into three cohorts: Screening cohort, High-Risk Screening, and Diagnostics cohort. Participants recruited for the study will be assigned to a dedicated cohort based on the reason of the visit.

There will be two visits for study participants, partially including study specific and routine procedures, who meet the inclusion criteria in the screening procedure.

The first trial visit (V1.1) will take place to provide the patient with detailed information on the study, its aims, the ThermoBreast procedure, and its risks. In- and exclusion criteria will be checked. Informed consent will be obtained. If the patient consents, the study specific ThermoBreast procedure (index test) and a study specific questionnaire regarding user experience will be performed. Moreover, the patient will undergo the routine first breast cancer screening round (screening cohort) or the routine first breast cancer diagnostics round (diagnostic cohort) according to national guidelines which serve as a reference test. In the screening cohort, the patient may undergo routine breast diagnostics following an irregular first screening round (V1.2) according to national guidelines.

The second trial visit (V2) serves as a follow-up visit for the reference test - no study specific interventions will be performed here. Patients will undergo routine breast cancer screening or diagnostics according to national guidelines which serve as a reference test. In the screening cohort, the patient may undergo routine breast diagnostics following an irregular second screening round (V2.2) according to national guidelines. No study specific interventions will be performed during this trial visit.

There will be no randomization within this study design. The findings of thermal screening will not be disclosed to patients and physicians, to avoid any anxiety or influence on the physicians' decision-making, as the proposed method is under study and development. The ThermoBreast system will only record the thermal imaging but will not automatically display any final assessment with respect to risk of breast cancer.

AI-based evaluation of dynamic breast thermography imaging (=ThermoBreast, index test) will serve as the outcome measure. The ThermoBreast evaluation will be performed independently of the routine breast diagnostic evaluation. Some baseline risk variables (e.g. patient age, hormonal status) may be included in the ThermoBreast evaluation. ThermoBreast will provide a risk score for invasive breast cancer on a per-patient basis (not per breast).

Routine breast diagnostics will serve as a reference test against which the ThermoBreast outcome will be compared. Depending on national guidelines and clinical scenarios, routine breast cancer diagnostics can consist of several routine procedures, including clinical examination, ultrasound, mammography, tomosynthesis, MRI, follow-up imaging, biopsy, surgical excision, and histopathologic evaluation. All procedures will be performed as indicated and specified by the respective, current national guidelines.

The AI-based evaluation will use state-of-the-art image analysis techniques. The algorithm will be trained on data acquired during the training phase of the trial. For the second 6 month validation phase of the trial, a data lock will ensure that outcomes with respect to the reference test (routine breast diagnostics) will not be available anymore for the team responsible for the ThermoBreast algorithm development.

A positive reference test is defined as histopathologic diagnosis of invasive breast cancer.

A negative reference test is defined as

* For the hypothesis without follow-up: a first study visit without biopsy indication (breast imaging BI-RADS 3,2 or 1), or a benign histopathologic evaluation.
* For the hypothesis with follow-up: two regular study visits (breast imaging BI-RADS 2 or 1), a regular follow-up imaging after an irregular screening/imaging finding (BI-RADS 3 followed by BI-RADS 2 or 1), or a benign histopathologic evaluation.

Analyses will be performed on a per-patient basis. In case of multiple breast masses per patient, the one with the highest risk of breast cancer or histopathological confirmed invasive breast cancer will be considered for the primary efficacy analysis

ELIGIBILITY:
Inclusion criteria

* Screening cohort

  * Female subjects aged 40 to 74 years old (inclusive) presenting for routine mammography/tomosynthesis breast cancer screening according to national/regional guidelines
  * Subjects who are willing to give written informed consent for study participation
  * Subjects who are able to understand the character and individual consequences of the clinical trial and who are ready to comply with the study related visits and procedures
* High-risk screening cohort

  * Female subjects aged 18 and above presenting for intensified high-risk breast cancer screening due to genetic predisposition or family history according to national/regional guidelines
  * Subjects who are willing to give written informed consent for study participation
  * Subjects who are able to understand the character and individual consequences of the clinical trial and who are ready to comply with the study related visits and procedures
* Diagnostics cohort

  * Female subjects aged 18 and above presenting for intensified aftercare after a history of breast cancer, patients with symptoms (nipple discharge, breast lump based on physician physical exam or self-breast exam), patients who were referred for additional examination (MRI, Ultrasound, fine-needle aspiration cytology (FNAC) or biopsy) based on suspicious imaging findings in either breast
  * Subjects who are willing to give written informed consent for study participation
  * Subjects who are able to understand the character and individual consequences of the clinical trial and ready to comply with the study related visits and procedures

Exclusion Criteria

• (High-risk) Screening and Diagnostics cohort

* Subjects who are pregnant or lactating
* Subjects who have undergone lumpectomy or mastectomy in the last 4 months at the time of study enrollment
* Subjects who have undergone cancer therapy (chemotherapy, start of hormonal therapy, radiotherapy, surgery) in the last 4 months at the time of study enrollment
* Subjects who have undergone a breast biopsy in the last 2 months at the time of study enrollment
* No subject will be allowed to enrol in this trial more than once.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28000 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity (true-positive rate) | up to 2 years of follow-up
  As our primary outcome we will use true-positive ThermoBreast results, i.e. detected invasive breast cancer by ThermoBreast (=index test) compared to histopathologically confirmed invasive breast cancer during routine breast cancer screening/imaging (=reference test). We will report this outcome as the true-positive rate (=TPR, rate of patients with non-detected invasive breast cancer by ThermoBreast compared to histopathologically confirmed invasive breast cancer during routine breast cancer screening/imaging) which is a commonly used and validated measure in diagnostic studies.
Specificity (true-negative rate) | up to 2 years of follow-up
  As a co-primary outcome we will measure the specificity of the ThermoBreast screening modality. The specificity will be defined as the rate of true-negative ThermoBreast results, i.e., the number of correctly identified absence of invasive breast cancer by ThermoBreast, when compared to the number of absence of histopathologically confirmed invasive breast cancer or regular follow-up imaging during routine breast cancer screening/imaging. This outcome will be reported as the true-negative rate (=TNR, rate of patients for whom ThermoBreast correctly identifies the absence of invasive breast cancer in alignment with the results from routine breast cancer screening/imaging).

SECONDARY OUTCOMES:
Cancer detection rate | up to 2 years of follow-up
  To evaluate the invasive breast cancer detection rate per 1000 women screened of ThermoBreast and compare it with other standard breast cancer screening and diagnostic modalities (ultrasound, mammography, MRI)
Detection rate of ductal carcinoma in situ (DCIS) | up to 2 years of follow-up
  Number of women with ThermoBreast screening-detected ductal carcinoma in situ (if the pT category of the TNM classification falls into the category pTis) divided by the number of all women screened.
Detection rate of tumor category pT1 | up to 2 years of follow-up
  Number of women with ThermoBreast screening-detected invasive breast cancers of the category pT1 divided by the number of all women screened. A screening-detected breast cancer is classified as breast cancer of tumor category pT1 if tumor size is ≤ 20 mm in greatest dimension and the respective pT subcategory of the pTNM classification is one of the following: pT1mic, pT1a, pT1b, pT1c, pT1.
Recall rate | up to 2 years of follow-up
  To evaluate the recall rate per 100 women screened of ThermoBreast and compare it with other standard breast cancer screening and diagnostic modalities (ultrasound, mammography, MRI)
Sensitivity | up to 2 years of follow-up
  To evaluate the sensitivity of ThermoBreast and compare it with other standard breast cancer screening and diagnostic modalities (ultrasound, mammography, MRI)
Specificity | up to 2 years of follow-up
  To evaluate the specificity of ThermoBreast and compare it with other standard breast cancer screening and diagnostic modalities (ultrasound, mammography, MRI)
Positive-predictive value | up to 2 years of follow-up
  To evaluate the positive-predictive value of ThermoBreast and compare it with other standard breast cancer screening and diagnostic modalities (ultrasound, mammography, MRI)
Negative-predictive value | up to 2 years of follow-up
  To evaluate the negative-predictive value of ThermoBreast and compare it with other standard breast cancer screening and diagnostic modalities (ultrasound, mammography, MRI)
Diagnostic performance in the three trial cohorts | up to 2 years of follow-up
  To compare the diagnostic performance of ThermoBreast with routine breast cancer screening and imaging rate within the three cohorts ( (1) screening cohort, (2) high-risk screening cohort (3) diagnostics cohort) in terms of sensitivity, specificity, negative-predictive value, positive predictive value, recall rate, and cancer detection rate
Proportion of breast quadrant localization | Screening visit
  Number of women with correct localization of breast masses by ThermoBreast (measured in breast quadrants: upper outer, upper inner, lower outer, lower inner) divided by all women with breast masses.
Proportion of correct histopathologic subtype identification | up to 2 years of follow-up
  Number of women with correct diagnosis of histopathologic subtype by ThermoBreast (invasive-ductal, invasive-lobular, medullary, tubular, papillary, metaplastic, in-situ) divided by all women with the respective histopathologic subtype.
Proportion of correct tumorbiologic subtype identification | up to 2 years of follow-up
  Number of women with correct diagnosis of tumorbiologic subtype by ThermoBreast (hormon receptor positive/ HER2neu negative, hormon receptor positive, HER2neu positive, hormon receptor negative/HER2neu positive, triple-negative breast cancer) divided by all women with the respective tumorbiologic subtype.
Proportion of correct axillary lymph node involvement identification | up to 2 years of follow-up
  The compare the diagnostic performance of ThermoBreast to axillary ultrasound in the detection of axillary lymph node metastasis in terms of sensitivity and specificity
Effect of hormonal status on diagnostic performance | up to 2 years of follow-up
  To compare the diagnostic performance of ThermoBreast and routine breast imaging modalities in women with pre-,peri-,and post-menopausal status in terms of sensitivity, specificity, negative-predictive value, positive predictive value, recall rate, and cancer detection rate
Effect of breast density on diagnostic performance | up to 2 years of follow-up
  To compare the diagnostic performance of ThermoBreast and routine breast imaging modalities in women with different breast densities (ACR A-D) in terms of sensitivity, specificity, negative-predictive value, positive predictive value, recall rate, and cancer detection rate.
Effect of ethnicity on diagnostic performance | up to 2 years of follow-up
  To compare the diagnostic performance of ThermoBreast and routine breast imaging modalities in women with different ethnicity in terms of sensitivity, specificity, negative-predictive value, positive predictive value, recall rate, and cancer detection rate
Timing of ThermoBreast | up to 2 years of follow-up
  To estimate the possibility of ThermoBreast to replace versus precede routine breast cancer screening/imaging as an additional imaging technique in terms of diagnostic performance
Screening time | Screening visit
  To estimate the possibility to reduce the screening time by evaluating the effect of screening duration on the performance of ThermoBreast
Cost-effectiveness | up to 2 years of follow-up
  To evaluate the cost-effectiveness of ThermoBreast for breast cancer screening and diagnosis. A cost per QALY analysis will be conducted.
Lived Experience | Screening visit
  The goal is to measure the difference between thermography and mammography by patients' self-assessment. Concretely, we will focus on the following areas: trust in the modality, perceived pain and discomfort, intention to use and willingness to pay. For trust and reliability, we are going to use the existing Likert scale made by Cahour and Forzy (2009). Perceived pain and comfort will be measured via the Likert scale made by indication of pain in the bodymap (van der Grinten, 1991) and the pain intensity scale (Jensen and Karoly, 1986). The willingness to pay question is based on van Helvoort-Postulart et al.'s study (2008). The results will be assessed by ANOVA and t-test by evaluating differences between thermography and mammography, as well as expectations before the test and the actual experience after the test.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Golatta, MD, Study Director — University Hospital Heidelberg; André Pfob, MD, Principal Investigator — University Hospital Heidelberg
Locations (1):
- Heidelberg University Hospital, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://thermobreast.eu/